CLINICAL TRIAL: NCT03264443
Title: Combined Training and Health Education for Hypertensive Elders: a Multicenter Randomized Clinical Trial
Brief Title: Hypertension Approaches in the Elderly: a Lifestyle Study
Acronym: HAEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Pelotas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0044; 17-0044 (Other Grant/Funding Number: FIPE/Hospital de Clínicas de Porto Alegre)
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Hypertension
Keywords: physical activity; exercise; aging; older
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health education (Active Comparator): Patients will receive weekly lectures on hypertension related topics during 12 weeks.
  Interventions: Behavioral: Health education
- Combined training (Experimental): Patients will complete 12 weeks of combined training (aerobic + strength exercise, 3x/week) in a pragmatic setup. In order to make the interventions more similar, contents of the health education arm will also be discussed with patients receiving this intervention.
  Interventions: Behavioral: Combined training

INTERVENTIONS:
Behavioral: Health education — Weekly group lectures (1h each) giving information on patient's best practices to manage hypertension.
  Arms: Health education
Behavioral: Combined training — Combined training (aerobic and strength exercises), in moderate intensities (perceived exertion controlled) performed 3x/week (1h) duration with a education component (10') based on the contents of the health intervention.
  Arms: Combined training

SUMMARY:
Two-center randomized, parallel, controlled trial which will compare a pragmatic combined training program with a health education program in 184 older adults with hypertension. This study will last 12 weeks with assessments conducted at baseline, previously to the group allocation, and after interventions. There is a set of secondary outcomes which show clinical importance to the elderly population and are possibly influenced by the tested intervention.

DETAILED DESCRIPTION:
The present protocol describes a randomized controlled trial that aims to evaluate blood pressure effects of a pragmatic combined training program, with low equipment needs, in comparison with a health education program. The sample is composed by 184 older adults, divided in two implementation centers. Randomization ratio will be 1:1 and interventions will last 12 weeks, with three weekly sessions for the exercise arm and one to the health education arm. In order to analyze the effects of interventions in a comprehensive way, a range of variables related to ambulatory blood pressure (primary outcome), physical fitness, vascular and autonomous function, together with emotional and cognitive aspects will be evaluated in a pre-post fashion. The study's hypothesis, as well as the sample size calculation and analysis plan, is based on a superiority expectation for the exercise program in comparison with the health education program, especially for the blood pressure control, functional capacity and quality of life. The present study was designed and will be conducted by a multidisciplinary staff and follows ethical and methodological recommendations for clinical trials. It is expected that this multicenter randomized trial will provide scientific evidences with a high applicability to the non-pharmacological management of hypertension in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension diagnosis (through ambulatory blood pressure monitoring or medication use)
* Verified ability to exercise
* Unaltered pharmacological plan within previous 4 weeks
* Willingness to participate in any of interventions

Exclusion Criteria:

* Inability or refusal to give written consent
* Myocardial infarction, revascularization proceedings, deep vein thrombosis
* Severe cardiovascular disease (class III or IV heart failure, uncontrolled arrhythmia, unstable angina, or use of implantable defibrillator
* Chronic pulmonary disease which requires the use of oxygen or steroidal therapy
* Incidence of cardiovascular event, hospitalization or other severe health-related event during the experimental period
* High alcohol consumption (over 14 doses per week)
* Renal disease needing dialysis
* Language, cognitive or hearing problems
* Plans of moving to another city during the study
* Living together with another person enrolled in the study
* Osteoarticular or muscular injuries or another health conditions which generate inability to carry on the interventions
* Progressive neurological disorders (Parkinson, multiple sclerosis, etc.)
* Cancer treatment in the past 2 years
* A medical report indicating exercise counterindication based cardiopulmonary exercise testing

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure | Change from baseline 24-hour systolic blood pressure at 12 weeks
  24h ambulatory blood pressure measured through automatic oscillometric device

SECONDARY OUTCOMES:
Walking distance | Change from baseline walking distance at 12 weeks
  Longest distance walked as assessed by the six-minute walk test
Lower limbs functional capacity | Change from baseline SPPB score at 12 weeks
  By using the Short Physical Performance Battery (SPPB), lower-limb mobility will be assess in the following sequence: static standing balance, walking speed and indirect muscle strength
Cardiorespiratory fitness | Change from baseline VO2peak at 12 weeks
  Oxygen consumption at peak (VO2peak) as assessed by maximal cardiopulmonary exercise testing
Geriatric Depression Symptoms | Change from baseline GDS-15 score at 12 weeks
  15-item depression symptoms scale (GDS-15)
Quality of life (QoL) | Change from baseline QoL score at 12 weeks
  World Health Organization Quality of Life questionnaire
Autonomic function | Change from baseline beat-to-beat blood pressure variability at 12 weeks
  Basal and during Stroop Color-Word Conflict Test beat-to-beat blood pressure variability
Endothelial function, early adaptation | Change from baseline FMD at 6 weeks
  Flow-mediated dilatation (FMD) assessed through high resolution ultrasonography
Endothelial function | Change from baseline FMD at 12 weeks
  Flow-mediated dilatation (FMD) assessed through high resolution ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie S Pinto, PhD, Study Director — Federal University of Pelotas; Daniel Umpierre, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Universidade Federal de Pelotas, Pelotas, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after will be shared after trial completion. Data usage will be under the PI's auspices, but restrictions or screenings will not be imposed upon data requests. ABPM data and any deemed relevant support information (sociodemographic, clinical history and allocated groups) will be shared if available.Details regarding the study's design and statistical plan can be obtained consulting the trial's protocol. Data on other outcomes could be requested contacting the PI. Data access will be available after all participants completed the study and will remain accessible for as long as deemed necessary by the study's committee. Data sets, variables' dictionary and statistical analysis description will be made available online upon registration and acceptance of the study team's data sharing terms and policy.
Time Frame: The individual participant dataset will become available at a public repository up to six months after the first study publication.
Access Criteria: A simple registration will grant access to study datasets. The website for these files is not defined at the time of registration.

REFERENCES:
- [Derived] Schaun GZ, Alberton CL, Gomes MLB, Santos LP, Bamman MM, Mendes GF, Hafele MS, Andrade LS, Alves L, DE Ataides VA, Carmona MA, Lazaro R, Botton CE, Umpierre D, Pinto SS, Wilhelm EN. Maximal Oxygen Uptake Is Underestimated during Incremental Testing in Hypertensive Older Adults: Findings from the HAEL Study. Med Sci Sports Exerc. 2021 Jul 1;53(7):1452-1459. doi: 10.1249/MSS.0000000000002598. PMID 33449605
- [Derived] Umpierre D, Santos LP, Botton CE, Wilhelm EN, Helal L, Schaun GZ, Ferreira GD, De Nardi AT, Pfeifer LO, da Silveira AD, Polanczyk CA, Mendes GF, Tanaka H, Alves L, Galliano L, Pescatello LS, Brizio ML, Bock PM, Campelo P, Moraes RS, Domingues MR, Schaan BD, Alberton CL, Pinto SS; The HAEL Study Group. The "Hypertension Approaches in the Elderly: a Lifestyle study" multicenter, randomized trial (HAEL Study): rationale and methodological protocol. BMC Public Health. 2019 May 29;19(1):657. doi: 10.1186/s12889-019-6970-3. PMID 31142294